CLINICAL TRIAL: NCT03069573
Title: Phenotypic Characterization of Pediatric Patients With Esophageal Eosinophilia and Biomarkers Investigation for the Diagnosis of Eosinophilic Esophagitis
Brief Title: Phenotypic Characterization and Biomarkers Investigation for Eosinophilic Esophagitis in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Cristina Palmer Barros, Professor, Federal University of Uberlandia
Other Study IDs: CAAE-36787714.0.0000.5152
Record Dates: First submitted 2017-02-19; First posted 2017-03-03 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Eosinophilic Esophagitis; Gastroesophageal Reflux
Keywords: Eosinophilic Esophagitis; Gastroesophageal Reflux; Diagnose; Biomarker
MeSH Terms: conditions — Eosinophilic Esophagitis; Gastroesophageal Reflux; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — blood, saliva, esophageal tissue, esophageal mucus
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Eosinophilic Esophagitis - EoE: Diagnosis of pediatric EoE under current guidelines.
- Gastroesophageal reflux disease - GERD: Diagnosis of pediatric GERD under current guidelines.
- Control: Exclusion diagnosis of EoE or GERD, with non specific gastrointestinal general complaints.

SUMMARY:
The purpose of this study is to find out some potential biomarkers for the Eosinophilic Esophagitis (EoE) in pediatric patients through the prospective clinical characterization and assessment of samples collected during the diagnostic process

DETAILED DESCRIPTION:
This study collects clinical information from pediatric patients between 0-18 years old who have been undergoing upper gastrointestinal endoscopy due to general complaints. The demographic, clinical symptoms, endoscopy, pH monitoring, and histology data are assessed during the diagnostic process. In the baseline endoscopy procedure samples (blood, saliva, esophageal tissue, and esophageal mucus) are taken. After diagnostic process of EoE and Gastroesophageal reflux disease (GERD) supported by International Guidelines the patients are divided into three groups - EoE, GERD, and Control.

The techniques are used for patients characterization and assessment:

1. Symptoms score: General symptom score and/or Pediatric Eosinophilic Esophagitis Symptom Score (PEESS v2.0) - translated and adapted version for Brazilian Portuguese
2. Endoscopic Score: Eosinophilic Esophagitis (EoE) Endoscopic Reference Score (EREFS)
3. Peak eosinophil count (PEC) and histological features description
4. Proteomic analyses
5. Microbiome analyses
6. Immunohistochemistry analyses

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients who are undergoing upper gastrointestinal endoscopy for diagnostic purpose

Exclusion Criteria:

* Pediatric patients who are undergoing upper gastrointestinal endoscopy for therapeutic procedures
* The presence of other eosinophilic diseases
* Patients have been taken corticosteroids and/or gastric acid secretion inhibition drugs for the last four weeks

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Consecutive pediatric patients undergoing esophagogastroduodenoscopy (due to general complaints) at a Tertiary Public Health Care Center
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Biomarkers for the diagnose of Pediatric Eosinophil Esophagitis | 2016 August - 2017 March and 2018 November-December
  Identify diagnostic biomarker, able to distinguish EoE patients from GERD patients and other nonspecific gastrointestinal complains

SECONDARY OUTCOMES:
Endoscopic features of EoE | 2017 January-March and 2018 November-December
  Evaluation of the EREFS 'ability (endoscopic reference score) to identify EoE patients and the inflammatory or fibrosis phenotype
Symptoms of active EoE | 2017 January-March and 2018 November-December
  Evaluation of the symptom score's ability to identify EoE patients in active disease
Histological features of EoE | 2017 January-March and 2018 November-December
  Evaluation of the histologic score's ability to identify EoE patients and the inflammatory or fibrosis phenotype

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Ricardo Goulart, Professor, Study Director — Federal University of Uberlandia; Cristina Palmer Barros, Professor, Principal Investigator — Federal University of Uberlandia
Locations (1):
- Federal University of Uberlandia, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liacouras CA, Furuta GT, Hirano I, Atkins D, Attwood SE, Bonis PA, Burks AW, Chehade M, Collins MH, Dellon ES, Dohil R, Falk GW, Gonsalves N, Gupta SK, Katzka DA, Lucendo AJ, Markowitz JE, Noel RJ, Odze RD, Putnam PE, Richter JE, Romero Y, Ruchelli E, Sampson HA, Schoepfer A, Shaheen NJ, Sicherer SH, Spechler S, Spergel JM, Straumann A, Wershil BK, Rothenberg ME, Aceves SS. Eosinophilic esophagitis: updated consensus recommendations for children and adults. J Allergy Clin Immunol. 2011 Jul;128(1):3-20.e6; quiz 21-2. doi: 10.1016/j.jaci.2011.02.040. Epub 2011 Apr 7. PMID 21477849
- [Background] Vandenplas Y, Rudolph CD, Di Lorenzo C, Hassall E, Liptak G, Mazur L, Sondheimer J, Staiano A, Thomson M, Veereman-Wauters G, Wenzl TG, North American Society for Pediatric Gastroenterology Hepatology and Nutrition, European Society for Pediatric Gastroenterology Hepatology and Nutrition. Pediatric gastroesophageal reflux clinical practice guidelines: joint recommendations of the North American Society for Pediatric Gastroenterology, Hepatology, and Nutrition (NASPGHAN) and the European Society for Pediatric Gastroenterology, Hepatology, and Nutrition (ESPGHAN). J Pediatr Gastroenterol Nutr. 2009 Oct;49(4):498-547. doi: 10.1097/MPG.0b013e3181b7f563. PMID 19745761
- [Background] Hirano I, Moy N, Heckman MG, Thomas CS, Gonsalves N, Achem SR. Endoscopic assessment of the oesophageal features of eosinophilic oesophagitis: validation of a novel classification and grading system. Gut. 2013 Apr;62(4):489-95. doi: 10.1136/gutjnl-2011-301817. Epub 2012 May 22. PMID 22619364
- [Background] Singla MB, Chehade M, Brizuela D, Maydonovitch CL, Chen YJ, Riffle ME, Achem SR, Moawad FJ. Early Comparison of Inflammatory vs. Fibrostenotic Phenotype in Eosinophilic Esophagitis in a Multicenter Longitudinal Study. Clin Transl Gastroenterol. 2015 Dec 17;6(12):e132. doi: 10.1038/ctg.2015.62. PMID 26680264
- [Background] Dohil R, Newbury R, Fox L, Bastian J, Aceves S. Oral viscous budesonide is effective in children with eosinophilic esophagitis in a randomized, placebo-controlled trial. Gastroenterology. 2010 Aug;139(2):418-29. doi: 10.1053/j.gastro.2010.05.001. Epub 2010 May 7. PMID 20457157
- [Background] Aceves SS, Newbury RO, Dohil MA, Bastian JF, Dohil R. A symptom scoring tool for identifying pediatric patients with eosinophilic esophagitis and correlating symptoms with inflammation. Ann Allergy Asthma Immunol. 2009 Nov;103(5):401-6. doi: 10.1016/S1081-1206(10)60359-6. PMID 19927538
- [Derived] de Souza TA, Carneiro AP, Narciso AS, Barros CP, Alves DA, Marson LB, Tunala T, de Alcantara TM, de Paiva Maia YC, Briza P, Ferreira F, Goulart LR. Eosinophilic esophagitis auxiliary diagnosis based on a peptide ligand to eosinophil cationic protein in esophageal mucus of pediatric patients. Sci Rep. 2022 Jul 18;12(1):12226. doi: 10.1038/s41598-022-16293-1. PMID 35851408